## **ClinicalTrials.gov Cover Page**

**Official Study Title:** What are the isokinetic strength and self-reported functional outcomes (ATRS) at 12 months after non-surgical management of Achilles tendon rupture using the SMART protocol?

**NCT Number:** [Add NCT number after PRS approval]

**Document:** Informed Consent Form

Version: 1

Date: 21 January 2026

Sponsor: Liverpool University Hospitals NHS Foundation Trust

Responsible Party: Chief Investigator Jeff Morton

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.

Version Number: 1 Date: 21/01/2026

| IRAS ID: 357432 |
|---------------------------------------------------|
| Centre Number: |
| Study Number: |
| Participant Identification Number for this trial: |



## **CONSENT FORM**

Title of Project: What are the isokinetic strength outcomes and self-reported functional outcomes (ATRS) at 12 months following non-surgical management of Achilles tendon rupture using the SMART protocol?

Name of Researcher: Raymond Healy

| | Please | e initial box |
|---|---|---|
| 1. | I confirm that I have read the information sheet dated (version) for the above study. I have had the opportunity to consider the information, ask questions and have had these answered satisfactorily. | |
| 2. | I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my medical care or legal rights being affected. | |
| 3. | I understand that relevant sections of my medical notes and data collected during the study, may be looked at by individuals from the research team, from regulatory authorities of from the NHS Trust, where it is relevant to my taking part in this research. I give permission for these individuals to have access to my records. | r 🗌 |
| 4. | I understand that the information collected about me will be used to support other research in the future, and may be shared anonymously with other researchers. | |
| 5. | I agree to my General Practitioner being informed of my participation in the study. | |
| 6. | I understand that the information held and maintained by-Liverpool University Hospitals NHS Foundation Trust may be used to help contact me or provide information about my health status. | |
| 7. | I agree to take part in the above study. | |

When completed: 1 for participant; 1 for researcher site file; 1 to be kept in medical notes.

Version Number: 1 Date: 21/01/2026

| Name of Participant | Date | Signature |
|---------------------|------|-----------|
| Name of Person | Date | Signature |
| seeking consent | | |